CLINICAL TRIAL: NCT00684918
Title: A Multicenter, Open-Label, 2-Stage, Phase II Study of Single-Agent Obatoclax Mesylate Administered For Three Consecutive Days Every 2 Weeks to Older Patients With Previously Untreated Acute Myeloid Leukemia (AML)
Brief Title: Study of Obatoclax in Previously Untreated Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gemin X (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM016
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: AML
Keywords: AML, obatoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — obatoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): In the Pilot Schedule portion of the study 3 hour vs 24 hour infusion schedules of obatoclax.
  Interventions: Drug: Obatoclax

INTERVENTIONS:
Drug: Obatoclax — A 3-hour IV infusion for 3 consecutive days or a 24-hour infusion for 3 consecutive days every 2 weeks for up to 6 cycles.
  Other Names: GX15-070MS

SUMMARY:
This protocol will evaluate the efficacy of obatoclax in older patients with previously untreated AML.

DETAILED DESCRIPTION:
The Pilot Safety portion of the study will evaluate the safety of obatoclax administered by a 3 hour infusion for 3 days in a row. The Pilot Schedule portion of the study will randomize 16 patients in to one of two cohorts: 1) patients receiving obatoclax administered by a 3 hour infusion for 3 days in a row or 2) patients receiving obatoclax administered by a 24 hour infusion for 3 days in a row. The schedule with the best overall efficacy and safety in the Pilot Schedule portion of the study will then be utilized in the Phase II portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed AML
* No prior chemotherapy for AML (with the exception that the patients enrolled in the Pilot Safety evaluation may have had 1 prior therapy)
* Age ≥70 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2
* Patients must have normal organ function as defined below:

  1. Total bilirubin < or = 2 mg/dL unless resulting from hemolysis,
  2. Aspartate transaminase (AST [SGOT])/alanine transaminase (ALT [SGPT]) < or = 2.5 x institutional ULN
  3. Creatinine within normal institutional limits, OR creatinine clearance > or = 50 mL/min/1.73 meters squared for patients with creatinine levels above institutional ULN

Exclusion Criteria:

* Patients who have received or are receiving any other investigational or commercial agents or therapies administered with the intent to treat their malignancy (with the exception that the patients enrolled in the pilot safety evaluation may have had 1 prior therapy)
* patients with history of allergic reactions attributed to components of the formulated product (PEG300 and polysorbate 20)
* patients with history of seizure disorders or central nervous system leukemia
* patients with uncontrolled, intercurrent illness including, but not limited to, symptomatic neurological illness; active, uncontrolled, systemic infection considered opportunistic, life-threatening, or clinically significant at the time of treatment; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; significant pulmonary disease or hypoxia; or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Determine the rate of morphologic CR after treatment in the obatoclax single-agent therapy in older patients with previously untreated AML. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean Viallet, MD, Study Director — Gemin X Pharmaceuticals
Locations (13):
- United States (12):
  - Northwestern University, Chicago, Illinois
  - The University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center Research Institute, Westwood, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Michigan State University - Breslin Cancer Center, Lansing, Michigan
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - Legacy Emanuel Hospital & Health Center, Portland, Oregon
  - Penn State Hershey Cancer Institute-Clinical Trials Office, Hershey, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Schimmer AD, Raza A, Carter TH, Claxton D, Erba H, DeAngelo DJ, Tallman MS, Goard C, Borthakur G. A multicenter phase I/II study of obatoclax mesylate administered as a 3- or 24-hour infusion in older patients with previously untreated acute myeloid leukemia. PLoS One. 2014 Oct 6;9(10):e108694. doi: 10.1371/journal.pone.0108694. eCollection 2014. PMID 25285531